CLINICAL TRIAL: NCT01684059
Title: Study the Effect of Oral Zinc Supplementation on Enzymes of Nitric Oxide Pathway
Status: Completed | Type: Observational
Sponsor: Babylon University (Other)
Collaborators: Ministry of Health, Iraq (Network)
Responsible Party: Principal Investigator, mahmoud hussein hadwan, phD, Babylon University
Other Study IDs: Babil-2
Record Dates: First submitted 2012-09-09; First posted 2012-09-12 (Estimated); Last update posted 2012-09-12 (Estimated); Status verified 2012-09

CONDITIONS: Asthenozoospermia
MeSH Terms: conditions — Asthenozoospermia | interventions — Zinc Sulfate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single group: Single group: each participant receive same intervention (zinc sulfate) throughout study (non-randomized)
  Interventions: Dietary Supplement: zinc sulfate

INTERVENTIONS:
Dietary Supplement: zinc sulfate — every participant took two capsules of zinc sulfate per day for three months (each one 220mg)

SUMMARY:
The ability of spermatozoa to produce reactive oxygen species (ROS) has been respected since the 1940's. Oxidative stress limits the functional competence of mammalian spermatozoa via lipid peroxidation, the induction of oxidative DNA damage and the formation of protein adducts. Nitric oxide (NO) is a free radical generated from the oxidation of L-arginine to L-citrulline by reduced nicotinamide adenine dinucleotide phosphate (NADPH)-dependent NO synthases. Several studies suggest that the overproduction of this free radical and the subsequent excessive exposure to oxidative conditions have a potential pathogenetic implication, which due to the reduction of sperm motility. The present study was conducted to study the effect of Zn supplementation on the levels of NO synthase and arginase in semen of patients with asthenozoospmia.

DETAILED DESCRIPTION:
Previous studies suggest that high concentrations of NO play an injurious consequence on spermatozoa kinetic characteristics. These studies reported that NO may react with superoxide or hydrogen peroxide, resulting in the production of peroxinitrite, hydroxyl radical, or singlet oxygen, which cause oxidation of sperm membrane lipids and thiol proteins. NO also may inhibit cellular respiration by nitro-sylation of heme in mitochondrial enzymes, aconitase, and glyceraldehyde phosphate dehydrogenase, leading to a reduction of adenosine triphosphate and that is due to loss of motility of spermatozoa.

ELIGIBILITY:
Inclusion Criteria:

* the presence of asthenozoospermia in the semen sample.

Exclusion Criteria:

* the absence of endocrinopathy,
* varicocele, and
* female factor infertility. Smokers and alcoholic men were excluded from the study because of their recognized high seminal ROS levels and decreased antioxidant levels

Ages: 27 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Study Population: this study includes 60 fertile male partners from couples who had consulted the infertility clinic of babil hospital of maternity (Hilla city/ IRAQ).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2011-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Nitric oxide synthase activity | at the end of three months

SECONDARY OUTCOMES:
Arginase activity | at the end of three months

CONTACTS AND LOCATIONS:
Overall Officials: mahmoud H. hadwan, phD, Principal Investigator — babylon university / Iraq; Lamia A. Almashhedy, phD, Study Chair — Babylon university/Iraq; abdulrrazaq S. Alsalman, phD, Study Director — Babylon university/Iraq
Locations (1):
- Babylon university/ college of science, Hillah, Hilla, Iraq

REFERENCES:
- [Derived] Hadwan MH, Almashhedy LA, Alsalman AR. Study of the effects of oral zinc supplementation on peroxynitrite levels, arginase activity and NO synthase activity in seminal plasma of Iraqi asthenospermic patients. Reprod Biol Endocrinol. 2014 Jan 3;12:1. doi: 10.1186/1477-7827-12-1. PMID 24383664